CLINICAL TRIAL: NCT00357448
Title: Phase I Dose Escalation Study of Intraperitoneal (I.P.) ONTAK® Administered to Patients With Advanced Stage Ovarian Cancer
Brief Title: Denileukin Diftitox Used in Treating Patients With Advanced Refractory Ovarian Cancer, Primary Peritoneal Carcinoma, or Epithelial Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6193; NCI-2010-00832; NCT00268801 (obsolete NCT alias)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mixed Epithelial Carcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Undifferentiated Adenocarcinoma; Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer; Stage III Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — denileukin diftitox; Injections, Intraperitoneal; Enzyme-Linked Immunosorbent Assay; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive intraperitoneal denileukin diftitox over at least 15 minutes on days 1-3. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: denileukin diftitox; Procedure: intraperitoneal administration; Other: laboratory biomarker analysis; Other: enzyme-linked immunosorbent assay; Other: flow cytometry

INTERVENTIONS:
Biological: denileukin diftitox — Given IP at 3 dose levels: 5mcg/kg of ONTAK, 15mcg/kg of ONTAK, or 25mcg/kg of ONTAK
  Other Names: DAB389 interleukin-2; DAB389 interleukin-2 immunotoxin; DAB389-IL2; DAB389IL-2; DAB389IL2; DABIL2
Procedure: intraperitoneal administration — After completion of I.P. normal saline infusion, the I.P. catheter will be capped and patients will be turned/rotated for 1 hour to help facilitate I.P. bathing w/ONTAK; patients will be turned/rotated every 15 minutes in 4 different positions for a total of 1 hour
Other: laboratory biomarker analysis — Correlative studies
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
Other: flow cytometry — Correlative studies

SUMMARY:
RATIONALE: Biological therapies, such as denileukin difitox, may stimulate the immune system in different ways and may prevent tumor cells from growing. PURPOSE: This phase I trial is studying the side effects and best dose of denileukin diftitox in treating patients with advanced refractory ovarian cancer, primary peritoneal carcinoma, or epithelial fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To estimate the maximum tolerated dose of intraperitoneal administration of ONTAK. SECONDARY OBJECTIVES: I. To evaluate the change in the number of Tregs in the peritoneum with the administration of ONTAK. II. To evaluate the change in the number of Tregs in the peripheral blood with the administration of ONTAK. III. To assess the clinical impact of ONTAK on tumor burden by serial measurements of CA-125. IV. To assess the level of circulating cytokines IL-2, IL-6, IL-10, TGF-beta2, and TNF-alpha in the peritoneum and peripheral blood before and after I.P. ONTAK. OUTLINE: This is a dose escalation study. Patients receive intraperitoneal denileukin diftitox over at least 15 minutes on days 1-3. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of denileukin diftitox until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. After the completion of study treatment, patients are followed up at 1 and 2 weeks, monthly for 3 months, and then at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of epithelial ovarian carcinoma, primary peritoneal carcinoma, or epithelial fallopian tube carcinoma
* Patients with the following histologic epithelial cell types are eligible: Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, transitional cell carcinoma, and mixed epithelial carcinoma
* Patients with advanced stage refractory ovarian carcinoma: patients unable to achieve first complete remission (CR) with first or second line chemotherapy OR patients with disease relapse after achieving second CR
* Patients must be 30 days out from last chemotherapy; previous chemotherapy must include a platinumbased regimen and paclitaxel (Taxol)
* Patients must have undergone primary debulking surgery
* Patients must have a peritoneal catheter suitable for I.P. infusion
* White blood cell count (WBC) > 3.0 THOU/ul
* Serum creatinine =< 2.5 mg/dL
* ALT =< 2.5 x upper limit of normal
* AST =< 2.5 x upper limit of normal
* Total bilirubin =< 2.0 x upper limit of normal
* Albumin >= 3.0 g/dL
* Subjects must have a Performance Status Score (Zubrod/SWOG Scale) =< 2
* Subjects must have recovered from major infections and/or surgical procedures and, in the opinion of the investigator, not have a significant active concurrent medical illness precluding protocol treatment
* Lymphocytes > 1.0 THOU/ul
* Platelets >= 100 THOU/ul

Exclusion Criteria:

* Prior treatment with ONTAK (DAB389IL-2) or DAB486IL-2
* Known history of hypersensitivity to diphtheria toxin or IL-2
* Moderate (symptomatic requiring the use of diuretics) or severe (symptomatic requiring paracentesis or other invasive intervention) ascites
* Active autoimmune disease
* Known history of pulmonary disease except controlled asthma
* Known history significant cardiac disease
* Concurrent malignancy requiring active treatment
* Clinical or radiological evidence of acute bowel obstruction within 30 days of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-04; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity profile as assessed by the Cancer Therapy Evaluation Program, Common Terminology Criteria for Adverse Events version 3.0 | From baseline
MTD | From baseline

SECONDARY OUTCOMES:
Efficacy of ONTAK defined as a 25% reduction in the number of Tregs in either the peripheral blood and/or in the peritoneal cavity | From baseline
Clinical impact on course of disease as assessed by serum CA-125 measurements | At baseline and at months 1, 2, 3, and 6
Changes in circulating cytokines IL-2, IL-6, IL-10, TGF-beta2, and TNF-alpha in the peripheral blood and at the site of disease as measured by ELISA | Pre- and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lupe Salazar, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Liao JB, Jejurikar NS, Hitchcock-Bernhardt KM, Gwin WR, Reichow JL, Dang Y, Childs JS, Coveler AL, Swensen RE, Goff BA, Disis ML, Salazar LG. Intraperitoneal immunotherapy with denileukin diftitox (ONTAK) in recurrent refractory ovarian cancer. Gynecol Oncol. 2024 Dec;191:74-79. doi: 10.1016/j.ygyno.2024.09.019. Epub 2024 Oct 2. PMID 39362046